CLINICAL TRIAL: NCT04368091
Title: XTOSI Pilot Study: Clinical Use and Safety of the Xtreme Touch (Magic Touch PTA) - Neo Sirolimus Coated PTA Balloon Catheter in the Treatment of Infrainguinal Peripheral Arterial Disease
Brief Title: Clinical Use and Safety of the Xtreme Touch (Magic Touch PTA)- Neo Sirolimus Coated PTA Balloon Catheter in the Treatment of Infrainguinal Peripheral Arterial Disease
Acronym: XTOSI
Status: Completed | Type: Observational
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: XTOSI Pilot Study
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Artery Disease; Atherosclerosis
Keywords: PAD; BTK; SFA; DCB; SCB
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All-comers, real-world registry: Subjects requiring infrainguinal revascularization with the Xtreme Touch - Neo (Magic Touch PTA)
  Interventions: Device: Xtreme Touch - Neo sirolimus coated PTA balloon catheter

INTERVENTIONS:
Device: Xtreme Touch - Neo sirolimus coated PTA balloon catheter — The Xtreme Touch (Magic Touch PTA) - Neo Sirolimus PTA Balloon Catheter is the world's first sirolimus coated PTA balloon. The purpose of the X-TOSI all-comers registry is to collect short and long-term clinical performance data on the Xtreme Touch (Magic Touch PTA) -Neo sirolimus PTA balloon catheter in the treatment of atherosclerotic disease in the infrainguinal arteries in an all-comers patient population in real world daily clinical practice.
  Other Names: Magic Touch PTA - Sirolimus drug coated balloon

SUMMARY:
This study postulates that the application of Sirolimus, an anti-proliferative agent that inhibits neointimal hyperplasia, via Sirolimus coated balloon (SCB) will be safe and will result in better arterial patency in infrainguinal peripheral arterial disease (PAD). The aim is to evaluate the efficacy (12 month freedom from clinically driven target lesion revascularisation) and safety (freedom from major adverse events) of sirolimus coated balloons in the treatment of infrainguinal PAD.

DETAILED DESCRIPTION:
It is imperative to have effective treatment strategies for PAD which can maintain the patency of arteries. The current standard of care for PAD is angioplasty which includes usage of drug coated balloons (DCB). Paclitaxel is the only anti-proliferative drug available in all currently available DCB technology. Sirolimus is another highly effective anti-proliferative drug of immense potential as demonstrated by superior results in Sirolimus drug eluting stents in coronary disease. The physical properties of Sirolimus have made it challenging for it to be similarly applied to DCB technology and it is only due to recent advances in nanotechnology that it is now possible to develop Sirolimus coated balloons (SCB), which is the study device used in this study. The study device allows delivery and deposition of sirolimus to the arterial wall. By applying this agent into lesions in peripheral arterial disease, this study aim to effectively reduce neointimal hyperplasia, and therefore prolong the patency of the artery and improve our limb salvage rates for PAD and CLI patients. Subjects will be followed up in the clinic at 6 month, 12 month, and 24 month post-intervention to assess primary and secondary outcome of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years or minimum age
* Subject must be willing to sign a Patient Data Release Form or Patient Informed Consent where applicable
* Lesion(s) in the infrainguinal arteries between 3 to 6mm which are suitable for endovascular treatment treated with the Xtreme Touch - Neo sirolimus PTA balloon catheter. For below the knee (BTK) arteries, lesions located in the proximal 200mm of the artery.

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Subject is currently participating in another investigational drug or device study that has not reached ist primary endpoint yet
* Subject is pregnant or planning to become pregnant during the course of the study
* Failure to achieve less than 30% residual stenosis in pre-existing lesion after plain balloon angioplasty
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from an all-comers patient population with all subjects requiring infrainguinal revascularization with the Xtreme Touch - Neo.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: Number of Patients with Primary patency | 6 months
  Defined as by duplex ultrasonography-derived peak systolic velocity ratio of < = 2.4
Safety: Number of Patients with Freedom from Major Adverse Events (MAE) defined as composite of | 6 months
  1. freedom from device- and procedure-related mortality, and major target limb amputation through to 30 days, and
  2. Freedom from clinically driven target lesion revascularization (TLR) within 6 months post-index procedure.

SECONDARY OUTCOMES:
Number of Patients with Freedom from clinically-driven TLR | 6, 12, and 24 months
  Freedom From Clinically Driven Target Lesion Revascularization
Number of Patients with Freedom from clinically-driven TVR | 6 and 24 months
  Freedom From Clinically Driven Target Vessel Revascularization
Number of Patients with Primary patency | 12 and 24 months
  Percentage of subjects with duplex ultrasound Clinical Primary Patency
Number of Patients with Freedom from MAE | 12 and 24 months
  b. A composite of freedom from device- and procedure-related mortality, and major target limb amputation
Number of Patients with Amputation-free survival | 6, 12 and 24 months
  Amputation-free survival of patients
Number of Patients with Improvement in Rutherford classification | 6, 12 and 24 months
  Improvement in Rutherford classification compared to the pre-procedure Rutherford classification
Number of Patients with Device success | Day 0
  Successful delivery, inflation, deflation, and retrieval of the Xtreme Touch - Neo balloon catheter.
Number of Patients with Technical success | Day 0
  Successful completion of the endovascular procedure and immediate morphological success with ≤ 50% residual diameter reduction of the treated lesion as determined by visual estimation
Number of Patients with Procedural success | Participants will be followed for the duration of hospital stay, an expected average of 1-2 days
  Participants will be followed for the duration of hospital stay, an expected average of 1-2 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Choke Tieng Chek, Principal Investigator — edward.choke.t.c@singhealth.com.sg
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacoppo D, Cassese S, Harada Y, Colleran R, Michel J, Fusaro M, Kastrati A, Byrne RA. Drug-Coated Balloon Versus Plain Balloon Angioplasty for the Treatment of Femoropopliteal Artery Disease: An Updated Systematic Review and Meta-Analysis of Randomized Clinical Trials. JACC Cardiovasc Interv. 2016 Aug 22;9(16):1731-42. doi: 10.1016/j.jcin.2016.06.008. PMID 27539695
- [Background] Clever YP, Peters D, Calisse J, Bettink S, Berg MC, Sperling C, Stoever M, Cremers B, Kelsch B, Bohm M, Speck U, Scheller B. Novel Sirolimus-Coated Balloon Catheter: In Vivo Evaluation in a Porcine Coronary Model. Circ Cardiovasc Interv. 2016 Apr;9(4):e003543. doi: 10.1161/CIRCINTERVENTIONS.115.003543. PMID 27069105
- [Background] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764